CLINICAL TRIAL: NCT01749787
Title: A Phase Ib Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Dose Escalation, Safety and Tolerability Study of PRTX-100 in Combination With Methotrexate or Leflunomide in Patients With Active Rheumatoid Arthritis
Brief Title: Safety Study of PRTX-100 With Methotrexate or Leflunomide to Treat Active Rheumatoid Arthritis
Acronym: SPARTA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protalex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRTX-100-104
Record Dates: First submitted 2012-12-06; First posted 2012-12-17 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: arthritis; rheumatoid; methotrexate; leflunomide
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Staphylococcal Protein A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1.5 mcg/kg (Experimental): PRTX-100 at 1.5 mcg/kg administered via infusion once per week for 5 weeks
  Interventions: Drug: PRTX-100 at 1.5 mcg/kg
- 3.0 mcg/kg (Experimental): PRTX-100 at 3.0 mcg/kg administered via infusion once per week for 5 weeks
  Interventions: Drug: PRTX-100 at 3.0 mcg/kg
- 6.0 mcg/kg (Experimental): PRTX-100 at 6.0 mcg/kg administered via infusion once per week for 5 weeks
  Interventions: Drug: PRTX-100 at 6.0 mcg/kg
- 12.0 mcg/kg (Experimental): PRTX-100 at 12.0 mcg/kg administered via infusion once per week for 5 weeks
  Interventions: Drug: PRTX-100 at 12.0 mcg/kg
- 240 mcg (Experimental): PRTX-100 at 240 mcg/dose administered via infusion once per week for 5 weeks then once every four weeks for 16 weeks thereafter.
  Interventions: Drug: PRTX-100 at 240 mcg
- Placebo (Placebo Comparator): Placebo administered via infusion once per week for 5 weeks
  Interventions: Drug: Placebo
- 420 mcg (Experimental): PRTX-100 at 420 mcg/dose administered via infusion once per week for 5 weeks then once every four weeks for 16 weeks thereafter.
  Interventions: Drug: PRTX-100 at 420 mcg

INTERVENTIONS:
Drug: PRTX-100 at 1.5 mcg/kg
  Other Names: Staphylococcal Protein A; SpA
  Arms: 1.5 mcg/kg
Drug: PRTX-100 at 3.0 mcg/kg
  Other Names: Staphylococcal Protein A; SpA
  Arms: 3.0 mcg/kg
Drug: PRTX-100 at 6.0 mcg/kg
  Other Names: Staphylococcal Protein A; SpA
  Arms: 6.0 mcg/kg
Drug: PRTX-100 at 12.0 mcg/kg
  Other Names: Staphylococcal Protein A; SpA
  Arms: 12.0 mcg/kg
Drug: PRTX-100 at 240 mcg
  Other Names: Staphylococcal Protein A; SpA
  Arms: 240 mcg
Drug: Placebo — Placebo administered via infusion once per week for 5 weeks
  Arms: Placebo
Drug: PRTX-100 at 420 mcg
  Other Names: Staphylococcal Protein A; SpA
  Arms: 420 mcg

SUMMARY:
The purpose of this study is to determine the safety and tolerability of PRTX-100 when various doses are given 5 times at weekly intervals to patients with active rheumatoid arthritis that are taking methotrexate or leflunomide. The drug is administered in a physician's office via an intravenous infusion. PRTX-100 may be effective in rheumatoid arthritis by suppressing the immune responses.

PRTX-100 is a highly-purified bacterial protein called Staphylococcal Protein A. In this study, cohorts of patients with active RA will receive sequentially higher doses of PRTX-100. There will be an inactive placebo cohort for comparison. Patients who do not attain low RA disease activity, by a commonly used measure, will leave the study at 3 months after their first dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Active RA with disease duration of not less than 6 months
* Concomitant stable methotrexate or leflunomide therapy

Exclusion Criteria:

* Diagnosis of any other inflammatory arthritis
* ACR Functional Classification of IV
* Significant systemic involvement secondary to RA (except for secondary Sjogren's syndrome)
* History of clincally significant hypogammaglobulinemia, common variable immunodeficiency, or humeral immunodeficientncy
* History of active tuberculosis, pro-thrombotic disorder, venous thrombosis requiring anti-coagulation, substance abuse, or serious psychiatric condition
* History of allergy or hypersensitivity to aspirin or non-steroidal cyclooxygenase inhibitors, Staphylococcal protein A
* History or presence of malignancy (except for surgically treated basal or squamous cell carcinoma of the skin at least 3 months prior to the start of study medication)
* Uncontrolled diabetes or Type 1 diabetes
* Unstable ischemic heart disease
* Serious active or recurrent infection, hepatic cirrhosis, or other medically unstable condition
* Systemic autoimmune diseases other than RA (such as systemic lupus erythematosus, scleroderma, inflammatory bowel disease, inflammatory myopathy)
* Positive for HIV, hepatitis B surface antigen, or hepatitis C antibody
* Pregnant or nursing females
* Inadequate hepatic, renal, or hematologic function
* Receipt of live vaccine within 5 weeks of start of study medication
* Concomitant administration of other biologic or non-biologic DMARDS, corticosteroids, or anti-CD20 antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Screening up to 53 Weeks
  Number, severity and attribution of relatedness of Adverse Events
Vital Signs and Physical Examinations | Screening up to 25 Weeks
  Change from baseline in blood pressure, heart rate, body temperature, and physical examination parameters
ECG | Screening, first dose, 5th dose, 9 weeks, and 25 weeks
  Change from baseline in heart rate, PR interval, QT/QTc interval and QRS duration
Clinical Laboratory Testing | Screening up to 25 weeks
  Change from baseline in blood chemistry, hematology, and urinalysis values

SECONDARY OUTCOMES:
Disease activity | Screening up to 53 weeks
  Number and percentage of patients attaining an ACR20, ACR50 and ACR70 response at Week 13. Change from baseline in CDAI, RAPID 3, and DAS28-CRP scores.
Immunogenicity | Prior to first dose, and at 4 weeks, 9 weeks, and 25 weeks
  Proportion of patients sero-positive and/or with titers > 512 at Week 4 and Week 9, the correlation between anti-product antibody and product clearance, and association between anti-product antibodies and adverse events.
Pharmacokinetics | Prior to first dose up to 72 hours after last dose of PRTX-100
  Plasma Cmax, AUC0-n, clearance and Vd.

CONTACTS AND LOCATIONS:
Overall Officials: William E Gannon, M.D., Study Director — Protalex, Inc.
Locations (8):
- United States (8):
  - Protalex Investigative Site, Los Angeles, California
  - Protalex Investigational Site, Sarasota, Florida
  - Protalex Investigational Site, Coeur d'Alene, Idaho
  - Protalex Investigational Site, Anderson, Indiana
  - Protalex Investigational Site, Albuquerque, New Mexico
  - Protalex Investigational Site, Salisbury, North Carolina
  - Protalex Investigational Site, Duncansville, Pennsylvania
  - Protalex Investigational Site, Allen, Texas